CLINICAL TRIAL: NCT03688763
Title: A Pilot Study of Digital Cognitive Behavioral Therapy for Veterans With Insomnia and Comorbid Psychopathology
Brief Title: A Pilot Study of Digital Cognitive Behavioral Therapy for Veterans
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID-19 related challenges in recruitment and conduct of study, the study was closed.
Sponsor: Palo Alto Veterans Institute for Research (Other)
Collaborators: Big Health Inc. (Industry)
Responsible Party: Principal Investigator, Shannon McCaslin, Clinical Psychologist, Palo Alto Veterans Institute for Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC0002ARG
Record Dates: First submitted 2018-04-03; First posted 2018-09-28 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Insomnia
Keywords: insomnia; anxiety; PTSD
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Anxiety Disorders; Stress Disorders, Post-Traumatic | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Digital CBTi administered (Other): Participants will receive 6 sessions of digitally administered CBTi using the Sleepio platform over the course of 12 weeks. Each session lasts on average 30-60 minutes, and is tailored to participant's progress and problems. During the treatment phase, between sessions, participants complete the Consensus Sleep Diary to track their progress.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia (CBT-i)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia (CBT-i) — CBT-i is an evidence-based treatment for insomnia. Participants will receive CBT-i via online program (Sleepio).

SUMMARY:
The proposed study is a multiple baseline design pilot study which seeks to evaluate the impact of digitally administered CBT-I, using the Sleepio platform, for the treatment of insomnia disorder among Veterans with co-morbid psychopathology. In addition, information related to acceptability and feasibility of the intervention among a Veteran sample will be obtained.

DETAILED DESCRIPTION:
Cognitive Behavioral Therapy for Insomnia (CBT-I) is considered the front-line intervention for individuals with insomnia and has recently been rolled-out throughout the Veterans Health Administration (VHA; Manber et al., 2012). CBT-I includes behavioral (sleep restriction, stimulus control, relaxation exercises), cognitive (cognitive restructuring, mindfulness exercise), and psychoeducation (sleep hygiene) components. While CBT-I has been demonstrated to be a highly efficacious and effective intervention, it is a specialized intervention that can be costly and is in limited supply based on the level of training required and number of providers available. For this reason, digital administration of CBT-I has been examined and research has demonstrated initial efficacy among community samples (Ritterband et al., 2009; Vincent et al., 2009; Espie et al., 2012), with one platform, Sleepio, demonstrating efficacy compared to a placebo intervention (Espie et al., 2012; Espie et al., 2014). For this reason, the current study will utilize the Sleepio platform which provides an interactive, customized and tailored delivery of CBT-I.

ELIGIBILITY:
Inclusion Criteria:

Participants must be:

* at least 18 years of age (no upper age limit)
* meet DSM-5 defined criteria for insomnia disorder
* be on a stable dose of any prescription medication (including sleep medication) for at least 2 weeks prior to the in-person screening assessment
* have comorbid psychopathology (i.e., symptoms of Posttraumatic Stress Disorder (PTSD), anxiety, and/or depression)

Exclusion Criteria:

* limited mental competency (not oriented to person, place, or time) and the inability to give informed, voluntary, or written consent to participate
* high risk for sleep apnea (STOP-Bang score >/= 3)
* current or previous diagnosis of sleep apnea that is untreated
* history of moderate or severe Traumatic Brain Injury
* current substance or alcohol use disorder, moderate to severe, in the past 3 months
* current bipolar disorder
* current or lifetime psychotic disorders
* seizure disorders
* moderate to high risk of suicide in the past month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2023-06-21 (Actual)

PRIMARY OUTCOMES:
Changes in the Insomnia Severity Index (ISI) | 0 weeks (baseline), 12 weeks (end of Intervention Phase), and 16 weeks (Follow-Up)
  The ISI is used to assess self-reported insomnia severity (Bastien et al., 2001). It is a 7-item self-report scale assessing sleep problem severity over the last two weeks, rated on a 5-point scale from 0 to 4; a higher score indicates higher severity. The ISI sums scores on the 7 items (1a, 1b, 1c, 2, 3, 4, 5) for a total score range of 0 to 28.
Changes in Consensus Sleep Diary (CSD) | 12 weeks (end of Intervention Phase) and 16 weeks (Follow-Up)
  The CSD (Carney et al., 2012) will be used to monitor self-reported sleep during the baseline phase, over the course of the digitally administered CBT-I intervention, and throughout follow-up. The CSD is a standardized sleep diary based on expert consensus and qualitative patient input.
Changes in Participant Perception of the Acceptability, Perceived Value, and Feasibility of using a Digital Modality to Treat Insomnia Symptoms | 12 weeks (end of Intervention Phase) and 16 weeks (Follow-Up)
  This unpublished measure requests information on the participants impressions of using digitally administered CBT-i. Questions ask about the following areas: 1) Use of the digitally administered intervention including general impressions and frequency of use, 2) Perceived value and helpfulness of the digitally administered intervention including which features of the program were perceived to be most useful and how the program impacted different aspects of insomnia and management of insomnia, 3) Impact on health (e.g., perceived impact on management of insomnia), 4) Potential enhancements (i.e. recommendations for improvements to the intervention).

SECONDARY OUTCOMES:
Changes in The Posttraumatic Checklist-5 (PCL-5) | 0 weeks (baseline), 12 weeks (end of Intervention Phase), and 16 weeks (Follow-Up)
  The PCL-5 is a self-report measure of PTSD symptom severity (Weathers et al., 2013). The PCL is a 20-item measure which asks respondents how much they had been bothered in the prior month by their most traumatic experience. Item responses range from 0 (not very much) to 4 (extremely) with a total score range is 0-80. DSM-5 symptom cluster scores sum item scores: Cluster B (items 1-5), C (6-7), D (8-14), and E (items 15-20).
Changes in The Patient Health Questionnaire: Depression Scale (PHQ-9) | 0 weeks (baseline), 12 weeks (end of Intervention Phase), and 16 weeks (Follow-Up)
  The PHQ-9 is a 9-item self-report scale assessing depression over the last two weeks (Kroenke et al., 2002). An additional item asking about global depression and interference with life activities is not included in the PHQ-9 score. Items are scored from 0 (not at all) to 3 (nearly every day), for a total score range of 0 to 27.
Changes in the Generalized Anxiety Disorder 7-Item Scale (GAD-7) | 0 weeks (baseline), 12 weeks (end of Intervention Phase), and 16 weeks (Follow-Up)
  The GAD-7 is a 7-item anxiety scale (Spitzer et al., 2006) assessing symptoms over the past two weeks. Item scores range from 0 (not at all) to 3 (nearly every day). Items are summed to yield a total score.
Changes in The Brief Inventory for Psychosocial Functioning (B-IPF) | 0 weeks (baseline), 12 weeks (end of Intervention Phase), and 16 weeks (Follow-Up)
  The B-IPF-7 is a 7-item measure scored from 0 (not at all) to 6 (very much) (Bovin et al., 2018). The total score is the mean of the sum of all 7 items. The B-IPF assesses social functioning, academic and occupational functioning, daily activities over the past 30 days.

CONTACTS AND LOCATIONS:
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No